CLINICAL TRIAL: NCT03402321
Title: Clinical Comparison of Alveogyl and Gelatin Sponge in the Management of Pain After Epithelialized Free Gingival Graft Harvesting: A Randomized Clinical Trial
Brief Title: Alveogyl and Gelatin Sponge in the Management of Pain After Epithelialized Free Gingival Graft Harvesting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karim ehab gerges (Other)
Responsible Party: Sponsor-Investigator, Karim ehab gerges, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1792013
Record Dates: First submitted 2017-12-27; First posted 2018-01-18 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pain, Procedural
Keywords: alveogyl, gelatin sponge, free gingival graft, palate, pain
MeSH Terms: conditions — Pain, Procedural; Pain | interventions — Vaginal Creams, Foams, and Jellies; butyl aminobenzoate, eugenol, iodoform, spearmint oil drug combinations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): Gelatin Sponge Sheet is a heamostatic agent act as a mechanical barrier to protect the palatal donor site
  Interventions: Drug: Gelatin Sponge Sheet
- intervention group (Experimental): alvogyl in a paste form with analgesic action to protect the palatal donor site and help to relief pain
  Interventions: Drug: Alvogyl

INTERVENTIONS:
Drug: Gelatin Sponge Sheet — sheets act as a mechanical barrier used to protect the denuded area of the palatal donor site
  Other Names: gel foam
  Arms: control group
Drug: Alvogyl — paste form with analgesic action to protect the palatal donor site and help to relief pain
  Other Names: Alveogyl
  Arms: intervention group

SUMMARY:
clinical comparison between alvogyl and gelatin sponge when used to protect the denuded area of the palatal donor site after free gingival graft in means of reducing pain and healing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for different periodontal and peri-implant plastic surgeries requiring palatal mucosal graft harvesting
2. Systemically healthy

Exclusion Criteria:

1. Severe gagging reflex
2. Smokers
3. Occlusal trauma at site of graft
4. Pregnancy
5. Psychiatric disorder
6. Patients allergic to the used agents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
pain score | 2 weeks
  recorded by the pain trough a Visual Analogue scale score (between 0 and 10. 0: no pain, 1: minimal pain,10: severe pain)

SECONDARY OUTCOMES:
healing | 4 weeks
  healing of the palatal mucosa using H2O2 Test this test is based on the principle that if the epithelium is discontinuous, then H2O2 diffuses into the CT, the enzyme catalase acts on H2O2to release water and oxygen. This is shown clinically by the production of bubbles on the wound. The area to be evaluated is then dried, and 3% H2O2 is sprinkled on the wound with a syringe, waiting for the appearance of bubbles, which will suggest that the surgical site is not completely epithelialized. Complete healing will be recorded as a dichotomous variable (yes/no).
bleeding | 2 weeks
  Questionaire, Binary (yes or no).
analgesic consumption | 2 weeks
  questionaure, Numerical, Amount of analgesics daily consumption

REFERENCES:
- [Derived] Ehab K, Abouldahab O, Hassan A, Fawzy El-Sayed KM. Alvogyl and absorbable gelatin sponge as palatal wound dressings following epithelialized free gingival graft harvest: a randomized clinical trial. Clin Oral Investig. 2020 Apr;24(4):1517-1525. doi: 10.1007/s00784-020-03254-z. Epub 2020 Mar 6. PMID 32144515